CLINICAL TRIAL: NCT05738798
Title: A Randomized Controlled Trial to Investigate the (Cost)Effectiveness of Oral Immunotherapy With Different Allergens in Young Children With an Established Food Allergy
Brief Title: Oral Immunotherapy in Young Children With Food Allergy
Acronym: ORKA-NL
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Deventer Ziekenhuis (Other)
Collaborators: Dutch National Health Care Institute (Other); University of Twente (Other); Utrecht University (Other)
Responsible Party: Principal Investigator, Ted Klok, Principal Investigator, Deventer Ziekenhuis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL81774.075.22
Record Dates: First submitted 2022-12-20; First posted 2023-02-22 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Food Allergy
Keywords: Oral immunotherapy; infants; food allergy
MeSH Terms: conditions — Food Hypersensitivity | interventions — Immunotherapy

STUDY DESIGN:
Intervention Model Description: Randomized open trial (no placebo involved)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral immunotherapy (Experimental): oral immunotherapy, maintenance phase with daily 300 mg allergenic protein during 1 year
  Interventions: Dietary Supplement: oral immunotherapy
- routine care (No Intervention): strictly avoidance of the specific allergenic food

INTERVENTIONS:
Dietary Supplement: oral immunotherapy — oral immunotherapy is performed by freely available, widely used food products, regularly part of a normal infant's diet such as peanut butter or boiled egg.
  Arms: oral immunotherapy

SUMMARY:
The goal of this clinical trial is to learn about oral immunotherapy in food allergic children < 30 months of age. The main question it aims to answer is: What is the clinical- and cost-effectiveness of early low-dose oral immunotherapy aimed at long-term tolerance induction. Participants will receive oral immunotherapy for 1 year with a maintenance dose of 300 mg allergenic protein and are compared with food allergic infants not receiving oral immunotherapy to compare with natural tolerance development.

DETAILED DESCRIPTION:
Primary objective: What is the clinical- and cost-effectiveness of early low-dose oral immunotherapy aimed at long-term tolerance induction in children under the age of 30 months with an established food allergy compared to routine care? Secondary objective: What is the effect of early low-dose oral immunotherapy in children under the age of 30 months with an established food allergy on (allergy specific) quality of life of parents and children compared to routine care? Study design: randomized controlled superiority trial Study population: Children between 9 and 30 months old with an IgE-mediated food allergy to peanut, tree nuts, cow's milk and/or hen's egg as proven by an oral food challenge. Intervention: 1-year low-dose oral immunotherapy (daily 300 mg allergenic protein) compared to strict avoidance in the control group.

Main study parameters/endpoints: Long-term tolerance as assessed by an exit oral food challenge at 4 weeks after discontinuation of the oral immunotherapy, combined with uncomplicated consumption of a full dose of the specific food at 6 months after discontinuation of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* An IgE-mediated food allergy to peanut, cashew, hazelnut, walnut, cow's milk and/or hen's egg as proven by sensitization to the specific allergen (sIgE > 0.35kU/l) and a positive oral food challenge.
* The fore-mentioned allergens are introduced into the diet of the child (the child is tolerant for the specific allergen(s)), or the child is diagnosed with a food allergy for the specific allergen(s).

Exclusion Criteria:

* (Suspected) eosinophilic oesophagitis
* Uncontrolled asthma/ viral wheeze.
* The inability of parents to follow instructions, recognize allergic reactions or administer emergency medication.
* Participation in any other intervention study at the time of the OIT study, with the exception of studies on guided early introduction of highly allergenic foods.

Ages: 9 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with sustained unresponsiveness to consumption of a specific allergenic food 4 weeks after stopping the 1-year oral immunotherapy (OIT) | Timing of the OFC: week 57 (52 weeks of OIT, followed by a 4-week allergenic food-free interval)
  Definition of sustained unresponsiveness: a participant who passed an oral food challenge (OFC) to 4.2 gram of the allergenic protein.
  Definition of the allergenic protein: the allergenic protein which induced an allergic response at an OFC at the start of the study, and was administered to the patient during the OIT (i.e. milk, egg, peanut, hazelnut, cashew or walnut).
Percentage of tolerant participants at week 78 | week 78 = 6 months after stop of the 1-year oral immunotherapy
  In children achieving sustained unresponsiveness (outcome 1), the allergen is introduced into the diet by parents at a regular base. Six months after discontinuation of the OIT, tolerance to the specific allergenic protein is assessed.
  Definition of tolerant: Percentage of children with uncomplicated (i.e. without any allergic symptoms) consumption at home of a full dose of the specific allergenic protein (e.g. a glass of milk or a sandwich with peanut butter).
Cost-effectiveness ratio at 18 months (week 78). | 18 months (week 78).
  Incremental cost-effectiveness ratio (ICER) at 18 months (week 78). Costs associated with oral immunotherapy will be measured in Euros. Effectiveness will be considered as percentage of tolerant participants at week 78.
Cost-utility ratio at 18 months (week 78). | 18 months (week 78): at the end of the study period.
  Incremental cost-utility ratio (ICUR) will be calculated for both groups using health-related quality of life (HRQoL) scores from the AQoL-6D (assessment of quality of life - 6 dimensions) and converted to utility scores and will be expressed in euros per QALY.

SECONDARY OUTCOMES:
Health related quality of life of children, during the 1-year OIT and six months after the therapy (week 78) | during oral immunotherapy (T=0, 26 weeks and 52 weeks), and 6 months after stopping the oral immunotherapy (78 weeks)
  Children's quality of life as measured by:
  - Food Allergy Quality of Life Questionnaire - parental form (FAQLQ-PF) This questionnaire consists of 14 questions to be answered on a 7-point Likert-scale. Minimum score is 0 points (no impact of food allergy on quality of life), maximum score is 84 (high impact of food allergy on quality of life)
Occurrence of Adverse Event(s) Related to Oral Immunotherapy up to 65 weeks study participation | during build-up (up to 3 months) and 1-year oral immunotherapy, total 65 weeks
  (Serious) adverse events related to oral immunotherapy
Levels of allergy-related immune parameters | at start of the therapy and after 6 and 12 months maintenance therapy
  Levels of allergen specific IgE and IgG4
adherence | during 1 year oral immunotherapy
  Rate of daily providing the oral immunotherapy
Health related quality of life of parents, during the 1-year OIT and six months after the therapy (week 78) | during oral immunotherapy (T=0, 26 weeks and 52 weeks), and 6 months after stopping the oral immunotherapy (78 weeks)
  Parental quality of life as measured by:
  - Food Allergy Quality of Life- Parental Burden (FAQL-PB) This questionnaire consists of 17 questions to be answered on a 7-point Likert-scale. Minimum score is 0 points (no parental burden), maximum score is 102 (severe parental burden)

CONTACTS AND LOCATIONS:
Overall Officials: Ted Klok, MD PhD, Principal Investigator — Deventer Ziekenhuis
Locations (4):
- Netherlands (4):
  - Deventer hospital, Deventer, Overijssel
  - Amsterdam UMC, location AMC, Amsterdam
  - Reinier de Graaf Gasthuis, Delft
  - Martini hospital, Groningen

IPD SHARING:
Plan to Share IPD: Yes
Data collected for this study will be stored in SPSS and Excel and analyzed in SPSS.
  Access to trial IPD can be requested after the study is completed by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact wetenschapsbureau@dz.nl
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 01-07-2025 - 01-07-2026
Access Criteria: Researchers wanting to use the data would have to contact the PIs with a research proposal and Statistical Analysis Plan (SAP).

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT05738798/Prot_SAP_001.pdf